CLINICAL TRIAL: NCT05522322
Title: Role of Disease - Severity Scoring Systems in Predicting Out Come Among COPD Patients Admitted at Assiut University Hospital
Brief Title: COPD Scoring Systems in ICU
Acronym: crosssectional
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebtesam Mohamed Thabet, resident doctor, Assiut University
Other Study IDs: C0PD scoring systems
Record Dates: First submitted 2022-08-28; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: COPD Scoring System
MeSH Terms: interventions — Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COPD scoring ststems in ICU — SAPS & APACH scoring systems in COPD ICU pts

SUMMARY:
The aim of our study was to assess the performance of APACHE II and SAPS II scoring methods in predicting out come among critically ill COPD patients admitted to the respiratory intensive care unit (RICU) at Assiut University Hospital

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a progressive and debilitating airway disease that results in a large burden, both medically and financially. It affects millions of people around the world and causes great rates of morbidity and mortality. This burden is anticipated to increase with an estimated 5.8 million deaths annually by 2030 [1].

A large proportion of patients with COPD usually require admission to the ICU and it may be helpful to recognize patients at the time of admission who are probable to have bad consequence, so that these patients can be managed violently [2 There are many ICU scoring models, and numerous new systems are being progressed to assess severity of illness in ICU patients. The use of scoring models particularly developed for patient evaluation at the time of ICU entry has decreased many troubles and helped therapy delineation.

Acute Physiology and Chronic Health Evaluation II (APACHE II) and Simplified Acute Physiology Score II (SAPS II) scoring systems are the two models that are greatly used by the majority of ICUs to forecast the clinical consequence [3

ELIGIBILITY:
Inclusion Criteria All patients involved have undergone full history with special stress on age, gender, special habits, and associated diseases. Information such as the patient's need for mechanical ventilation as well as the duration of lodging in the ICU was entered. Routine laboratory variables were also registered. Patients were followed up until their outcome was determined. The outcome was decided according to the mortality within the ICU and recorded as survivors and nonsurvivors. Scores of

APACHE II and SAPS II were calculated:

-

Exclusion Criteria:

* Excluded from this study were COPD patients admitted to the ICU because of any other underlying problem such as those with acute cardiac situation, patients with respiratory failure due to other diseases along with COPD, patients who lasted less than 24 h in the ICU, and those who died before the completion of data collection.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Role of disease - severity scoring systems in predicting out come among COPD patients admitted at Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
COPD scorng systems in ICU | Baseline
  Role of disease - severity scoring systems in predicting out come among COPD patients admitted at Assiut University Hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Ebtesam, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Retraction. J Thromb Haemost. 2021 Aug;19(8):2096. doi: 10.1111/jth.15210. Epub 2021 Jan 1. PMID 33314547